CLINICAL TRIAL: NCT04086862
Title: Effect of Ultrasound Therapy on Bilateral Masseter Myalgia: Comparison of 1 Megahertz Versus 3 Megahertz
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, W.D.McCall, Jr., Professor, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Study00001683
Record Dates: First submitted 2019-09-10; First posted 2019-09-12 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Adult Females; Bilateral Masseter Myalgia
Keywords: temporomandibular disorders; masseter myalgia; adult female
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Ultrasonic Therapy

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to double-blind treatment with 1 MHz or 3 MHz therapeutic ultrasound.
Who Masked: Participant, Care Provider
Masking Description: The frequency setting on the ultrasound machine will be set and known only to the principal investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The 1 MHz group (Active Comparator): The 1 MHz group will receive therapeutic ultrasound at the 1 MHz setting.
  Interventions: Procedure: Therapeutic ultrasound
- The 3 MHz group (Experimental): The 3 MHz group will receive therapeutic ultrasound at the 3 MHz setting.
  Interventions: Procedure: Therapeutic ultrasound

INTERVENTIONS:
Procedure: Therapeutic ultrasound — A commercially available ultrasound machine will provide 5 minutes of ultrasound at 0.4 watt/cm^2 and 100% duty cycle sequentially to each masseter muscle.

SUMMARY:
Temporomandibular disorders (TMD) are a group of musculoskeletal and neuromuscular conditions that involve the temporomandibular joints, the masticatory muscles, and all associated tissues. These disorders are characterized by regional pain and limitation of mandibular range of motion. Pain-related TMD affects approximately 5% to 12% of the population and can affect individual's quality of life. The incidence is about 4 percent. Therapeutic ultrasound is a type of physical therapy that delivers energy via propagation of ultrasonic waves. One gap in knowledge is whether 1 megahertz (MHz) treating frequency has the same efficacy as treating with 3 MHz. This research proposes to test that.

DETAILED DESCRIPTION:
See brief summary.

ELIGIBILITY:
Inclusion Criteria:

* Adult females
* Bilateral myalgia based on Diagnostic Criteria for TMD (DC-TMD) criteria
* An average pain of 5 or more on a 0 to 10 scale over the last 30 days.

Exclusion Criteria:

* A history or diagnosis of systemic musculoskeletal disorders or rheumatologic diseases (e.g. fibromyalgia, muscular atrophy).
* Certain conditions such as neoplasms or fractures.
* Neuropathies or neurological disorders.
* Currently taking muscle relaxants or analgesics.
* Undergone any form of physical therapy within the last 60 days.
* Severe bruxism requiring mouth-guard treatment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-10-24 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2021-03-20 (Actual)

PRIMARY OUTCOMES:
Reduction in masseter pain by visual analog pain scale. | Baseline to fifth week.
  Reduction in masseter pain as measured on a visual analog scale (VAS). The VAS runs from 0 (no pain at all) to 100 (worst pain imaginable).
Reduction in masseter pain by pressure pain threshold. | Baseline to fifth week.
  Reduction in masseter pain as measured with the pressure pain threshold (VAS). The VAS runs from 0 (no pain at all) to 100 (worst pain imaginable)..

CONTACTS AND LOCATIONS:
Overall Officials: W. D. McCall, Ph.D., Principal Investigator — State University of New York at Buffalo
Locations (1):
- School of Dental Medicine, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No
De-identified data may be shared after analysis completed.